CLINICAL TRIAL: NCT01780376
Title: Latency of Whole-Body Vibration Induced Reflex Muscle Activity
Brief Title: Latency of Vibration-Induced Reflex Muscle Activity
Acronym: LVIRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEAH FTR-8
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Effects of Vibration
Keywords: whole-body vibration; latency; reflex response; muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WBV group (Experimental): whole-body vibration (WBV) group
  Interventions: Procedure: whole-body vibration (WBV)

INTERVENTIONS:
Procedure: whole-body vibration (WBV) — whole-body vibration (4 mm amplitude, 25,30,35,40,45,50 Hz)
  Other Names: Cyclic mechanical loading

SUMMARY:
Whole Body Vibration (WBV) applies thrust force in opposite direction to gravity to body.This mechanical stimulation induces reflex muscular activity. Tonic vibration reflex (TVR) is most commonly cited mechanism to explain WBV-induced reflex muscular activity (WBV-IRMA), although there is no conclusive evidence that TVR occurs. The bone myoregulation reflex is another neurologic mechanism used to explain the effects of vibration on muscular performance.

Investigators hypothesized that latency of WBV-IRMA is different from latency of TVR. Primary aim of this study is to determine latency of WBV-IRMA. Secondary aim is to investigate whether WBV-IRMA is explained with TVR.

Twenty healthy young adult men are planned to include in this study. Participants will stand upright with their knees locked during WBV. PowerPlate Pro5 will be used for WBV. WBV with high amplitude at 25,30,35,40,45 and 50 Hz will be applied. Surface electrodes will be placed on both the soleus muscles. To measure TVR latency, piezo-electric accelerometer will be placed on the achilles tendon and this achilles tendon will be stimulated with spring based mechanical reflex hammer. Our pilot study was showed that motor unit potentials (MUAP) occurred in a 1:1 response with vibration. After confirmation of this finding, WBV-IRMA latency will be measured in the present study. To measure WBV-IRMA latency, piezo-electric force sensor will be placed between heel and WBV platform. Exact moment of initial strike of heel when thrust force expressed by WBV begin to be transferred to body will be determined. The time between moment of the initial strike and corresponding MUAP is defined as "WBV-IRMA latency". Piezo-electric stretch sensor will be placed between knee and malleol to simulate muscle spindle. The reflex muscle activity of soleus muscles will be measured by PowerLab (data acquisition system, ADInstruments, Australia) device.

This project is planed to be completed in 1 months.

DETAILED DESCRIPTION:
Whole-body vibration (WBV), as a method of exercise training, is becoming increasingly popular in physical therapy, rehabilitation, and professional sports, and is increasingly used in beauty and wellness applications due to its beneficial effects on the neuromusculoskeletal system. These benefits include improved strength, power, flexibility, jump height, and balance. However, little is known about the physiological mechanisms underlying the effects of WBV on muscular performance, although the presence of reflex muscle activity during WBV has been shown. Tonic vibration reflex is the most commonly cited mechanism to explain the effects of WBV on muscular performance, although there is no conclusive evidence that TVR occurs. Studies have reported that direct vibration applied to a muscle or tendon stimulates muscle spindles, thereby causing a tonic vibration reflex to occur. As highlighted by these studies, muscle spindle discharges are sent to the spinal cord through Group Ia afferents during muscle or tendon vibration. There, they activate motoneurones that cause the muscle to contract. However, it has been reported that the sensitivity of the muscle spindle decreases or does not increase and that presynaptic inhibition occurs in Group Ia afferent fibers with vibration.

The bone myoregulation reflex (BMR) is another neurologic mechanism used to explain the effects of vibration on muscular performance. BMR is a reflex mechanism in which osteocytes exposed to cyclic mechanical loading induce muscle activity. Osteocytes embedded in the bone matrix are interconnected by numerous dendritic processes, forming a wide, mechanosensitive cellular network. Osteocytes exposed to cyclic mechanical loading send mechanical input signals to the central nervous system, influencing the neuronal regulation of muscle activity.

Investigators hypothesized that latency of WBV-IRMA is different from latency of TVR. Primary aim of this study is to determine latency of WBV-IRMA. Secondary aim is to investigate whether WBV-IRMA is explained with TVR.

Twenty healthy young adult men are planned to include in this study. Participants will stand upright with their knees locked during WBV. PowerPlate Pro5 will be used for WBV. WBV with high amplitude at 25,30,35,40,45 and 50 Hz will be applied. Surface electrodes will be placed on both the soleus muscles. To measure TVR latency, piezo-electric accelerometer will be placed on the achilles tendon and this achilles tendon will be stimulated with spring based mechanical reflex hammer. Our pilot study was showed that motor unit potentials (MUAP) occurred in a 1:1 response with vibration. After confirmation of this finding, WBV-IRMA latency will be measured in the present study. To measure WBV-IRMA latency, piezo-electric force sensor will be placed between heel and WBV platform. Exact moment of initial strike of heel when thrust force expressed by WBV begin to be transferred to body will be determined. The time between moment of the initial strike and corresponding MUAP is defined as "WBV-IRMA latency". Piezo-electric stretch sensor will be placed between knee and malleol to simulate muscle spindle. The reflex muscle activity of soleus muscles will be measured by PowerLab (data acquisition system, ADInstruments, Australia) device.

This project is planed to be completed in 1 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Men with ages varying between 20 and 45 years
* Right-handed men

Exclusion Criteria:

* Bone, muscle/tendon, joint, vascular, dermatologic diseases in lower extremities and spine
* Medication that could affect the musculoskeletal system
* Postural abnormalities (scoliosis, kyphosis, etc)
* Systemic diseases

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
latency of reflex muscle activity | 1 month
  Whole-body vibration induced reflex muscle activity latency

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Bagcilar Training & Research Hospital; MUHARREM CIDEM, MD, Principal Investigator — Bagcilar Training & Research Hospital; HALIL I CAKAR, PhD, Principal Investigator — Fatih University Biomedical Engineering Instıtute
Locations (1):
- Bagcilar TRH, Istanbul, Turkey (Türkiye)